CLINICAL TRIAL: NCT02579525
Title: Targeted Tissue Perfusion Versus Macrocirculatory-guided Standard Care in Patients With Septic Shock [TARTARE-2S]- A Multicentre Randomized Controlled Trial
Brief Title: Targeted Tissue Perfusion Versus Macrocirculatory-guided Standard Care in Patients With Septic Shock
Acronym: TARTARE-2S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Ville Pettilä, Professor of Intensive Care Medicine, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TARTARE-2S-01
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Shock; Septic; Critical Illness
Keywords: septic shock; tissue perfusion; macrocirculatory; mean arterial pressure; vasopressor use; days alive free of organ support
MeSH Terms: conditions — Shock, Septic; Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted tissue perfusion guidance (TTP) (Experimental): TTP-guidance based on clinical signs of peripheral perfusion.
  Interventions: Other: Hemodynamical treatment TTP
- Macrocirculatory - guidance (MCG) (Active Comparator): MCG-guidance based on recommended macrocirculatory parameters.
  Interventions: Other: Hemodynamical treatment MCG

INTERVENTIONS:
Other: Hemodynamical treatment TTP — Based on capillary refilling time, peripheral temperature, mottling, diuresis, MAP safety limit monitoring
  Arms: Targeted tissue perfusion guidance (TTP)
Other: Hemodynamical treatment MCG — Based on MAP, CVP, urine output monitoring
  Arms: Macrocirculatory - guidance (MCG)

SUMMARY:
Background: The recommended monitoring and target levels in septic shock (SSC Guidelines 2012) including mean arterial pressure (MAP) target are not based on robust clinical data.

Objective: To test, if in patients with septic shock, tissue perfusion guided (TPG) treatment strategy leads to a faster resolution of hypoperfusion than the macrocirculatory target guided standard care.

Design: A prospective phase II two-parallel-group open-label randomized controlled trial

Interventions:

1. Intervention group- Targeted tissue perfusion guided (TTP) - care.
2. Control group - Macrocirculatory - guided (MCG) care.

Randomization: 1:1 stratified according to the site and presence or absence of known hypertension.

Trial size: 200 randomised patients in 4 ICUs.

DETAILED DESCRIPTION:
Study hypothesis: Targeting at clinical tissue perfusion (in the TTP arm) will decrease the use and untoward effects of vasopressors, and result in more days alive in 30-days without vasopressor or inotropic support and without lactatemia, in comparison with standard clinical care with preference of macrocirculatory targets (MCG arm).

Intervention group - Targeted tissue perfusion (TTP) care:

Primary targets /registration period

1. capillary refill time (CRT) / <3 sec/ every hour
2. skin mottling / absent / every hour
3. arterial lactate / <2.0 mmol/l/ per 2hr
4. peripheral temperature/ warm /every hour
5. urine output/ ≥0.5 mL/kg per hour/ every hour
6. mean arterial pressure (MAP) 50-65 mmHg (minimum as a safety limit)/ continuous

   * if previous hypertension 65- 70 mmHg
   * if oliguria 2-hour trial 75-80 mmHg (If diuresis better, continue 2hr and re-evaluate) Secondary target
7. Continuous mixed venous saturation (SvO2) >65%, if available

Control group - Macrocirculatory targets guided (MCG) standard care Primary targets

1. Mean arterial pressure (MAP) 65-75 mmHg /continuous

   ** if previous hypertension 75-80 mmHg

   *** if oliguria < 0.3 ml/kg, 2-hour trial 85-90 mmHg (If diuresis better, continue 2hr and re-evaluate)
2. Central venous pressure (CVP)/hourly, Adequate fluid therapy is indicated to restore clinical hypovolemia up to the recommended CVP-level of 8-12 mmHg, if needed
3. Urine output ≥ 0.5 mL/kg/h/ hourly Secondary target
4. Continuous SvO2 >65%, if available

ELIGIBILITY:
Inclusion Criteria:

* Septic shock defined as

  1. Septic infection AND
  2. systemic mean blood pressure > 65 mmHg requiring any dose of vasopressors (norepinephrine, vasopressin) despite adequate fluid resuscitation (minimum of 20 ml/kg crystalloids) AND
  3. Elevated lactate ≥ 3.0 mmol/L with suspected hypoperfusion

Exclusion Criteria:

* aged less than 18 or over 80 years
* any other probable condition than sepsis affecting or expected to affect the central nervous system including post cardiac arrest
* present or suspected myocardial ischemia
* acute pulmonary embolism
* terminal illness and not considered for full intensive care support
* use of extra-corporeal membrane oxygenation (ECMO)
* known liver disease - Child-Pugh -Class B or C
* confirmed chronic kidney disease known on admission
* known to be pregnant or lactating
* more than 4 hours from fulfilled inclusion criteria to randomization
* another probable cause of hyperlactatemia
* patients transferred from another ICU
* patients with active haematological malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Days alive in 30 days- without vasopressors/ inotropes or hyperlactatemia | 30 days
  • Days alive in 30 days with normal arterial blood lactate ( first confirmed value of < 2 mmol/L) AND without any inotropic or vasopressor agent

SECONDARY OUTCOMES:
Time to normalization of arterial blood lactate | 30 days
Days alive with normal arterial blood lactate in 30 days | 30 days
Days alive without any inotropic or vasopressor agent in 30 days | 30 days
Days alive without renal replacement therapy (RRT) in 30 days | 30 days
Days alive without mechanical ventilation in 30 days | 30 days
Days alive without any organ support (mechanical ventilation, renal-replacement therapy, vasopressor/ inotropic agents) in 30 days | 30 days
New acute kidney injury (AKI) (Kdigo stages I-III) | 30 days
Days alive outside hospital in 90 days | 90 days
Total amount of norepinephrine given up to day 5 | 5 days
Number/ total number of the following adverse reactions | 30 days
  ventricular tachycardia/ fibrillation , atrial fibrillation , myocardial infarction , skin necrosis , stroke , secondary bowel ischemia, limb ischemia, numbers of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ville Pettilä, Prof, Principal Investigator — Helsinki University Hospital/ Bern University Hospital; Stephan Jakob, Prof, Dr, Principal Investigator — Bern University Hospital
Locations (2):
- Helsinki University Hospital, Helsinki, Finland
- Inselspital, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Varis E, Pettila V, Poukkanen M, Jakob SM, Karlsson S, Perner A, Takala J, Wilkman E; FINNAKI Study Group. Evolution of Blood Lactate and 90-Day Mortality in Septic Shock. A Post Hoc Analysis of the FINNAKI Study. Shock. 2017 May;47(5):574-581. doi: 10.1097/SHK.0000000000000772. PMID 27755509
- [Background] Pettila V, Merz T, Wilkman E, Perner A, Karlsson S, Lange T, Hastbacka J, Hjortrup PB, Kuitunen A, Jakob SM, Takala J. Targeted tissue perfusion versus macrocirculation-guided standard care in patients with septic shock (TARTARE-2S): study protocol and statistical analysis plan for a randomized controlled trial. Trials. 2016 Aug 2;17:384. doi: 10.1186/s13063-016-1515-x. PMID 27484695